CLINICAL TRIAL: NCT02804854
Title: Sensing Using Neutrophil Activation Probe on the Intensive Therapy Unit
Acronym: SNAP-IT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: Medical Research Council (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AC16025
Record Dates: First submitted 2016-06-02; First posted 2016-06-17 (Estimated); Last update posted 2022-11-04 (Actual); Status verified 2016-12

CONDITIONS: Lung Disease
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Patients in ICU (Experimental): Delivery of Neutrophil Activation Probe (NAP) (80mcgs) to ventilated patients up to three times.
  Interventions: Drug: Neutrophil Activation Probe (NAP)

INTERVENTIONS:
Drug: Neutrophil Activation Probe (NAP) — Delivery of NAP by direct pulmonary administration followed by fibreoptic confocal microendoscopy. A total of 240 mcg (±25%) in three divided doses of 80 mcg (±25%).

SUMMARY:
Critically ill patients often succumb to acute respiratory disease (rapidly developing disease affecting the lungs). The lungs are the commonest organ to fail and require support in the intensive care environment. However, no accurate methods exist that can be used at the bedside to tell what is causing deterioration in a person's lungs. There are various examples of acute respiratory diseases that can occur as a result of numerous different causes, have a high risk of death and cannot be treated easily with drugs. When trying to accurately diagnose and classify these lung diseases there is a risk that the type of respiratory disease is misdiagnosed, missed or the level of severity is not captured. By using the field of optical molecular imaging and employing novel techniques and technologies, the investigators hope to demonstrate here that a bespoke chemical probe administered in micro doses (tiny doses) directly into the distal lung can rapidly and accurately detect activated neutrophils (cells of the immune system that are implicated in the development of these severe conditions), and so work towards a bedside test which could be used to diagnose, monitor and classify the disease in patients who are critically ill in the future. The population for this study are in intensive care where patients are normally intubated (have a breathing tube) due to the severity of their illness, this may be because of respiratory problems or respiratory problems can rapidly develop. Participants will have the chemical probe administered into their lungs and pictures taken through the tube already in place. As this probe lights up when it comes into contact with neutrophils the investigators will be able to tell if neutrophils are present. This will inform a larger study in which it's hoped that the method can be used to inform clinical decisions. The first procedure will take place within two days of initiation of mechanical ventilation and the direct contact with the study team will be completed within nine days.

ELIGIBILITY:
Inclusion Criteria:

For all participants:

* Participants aged 16 years or over
* Participants who are predicted to require intubation for more than two calendar days, with this assessment made by a clinician (Registrar or Consultant in Intensive Care) who is independent of the study team.
* Participants who have undergone chest radiological imaging within the preceding 48 hours prior to enrolment.
* Participants who can undergo study bronchoscopy within the initial time period (C.D. 0-2) of first intubation in their present hospital admission (as determined by the absence of exclusion criteria for bronchoscopy laid out below).

For BAL subset (up to a total of 10 participants)

* Permission given to undertake a BAL by independent attending consultant
* CONTROL BAL (n=5)

  o Absence of pulmonary infiltrates on the aforementioned chest radiological imaging
* ABNORMAL BAL (n=5)

  * Pulmonary infiltrate on chest radiological imaging
  * Suspicion of community acquired pneumonia or ventilator associated pneumonia as determined by the clinical care team.

Exclusion Criteria:

For enrolment into the study:

* Absence of consent from the participant or their personal or professional legal representative
* Documented history of allergy to fluorescein
* Pregnancy Prior to each bronchoscopy (as assessed within 24 hours of the start of the procedure)
* Investigator not available to perform bronchoscopy with NAP/FE within the pre-specified time
* Treatment withdrawal documented to take place within the next 24 hours
* Presence of pneumothorax or intercostal chest drain
* Refusal by the patient's attending intensive care consultant

Prior to each study blood sampling • Haemoglobin (Hb) < 6.5 g/dL.

Prior to each BAL

• Refusal to permit BAL by the participants attending consultant

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2016-12; Primary Completion 2022-07 (Actual); Study Completion 2022-07 (Actual)

PRIMARY OUTCOMES:
Reproducibility of NAP signal | Length of the study - two years
  The reliability of the NAP/FE procedure as determined by the reproducibility of NAP signal during multiple transbronchial passes of the same segment in the same patient, averaged over the entire enrolled population.
Discriminant ability of NAP signal in normal or abnormal lung segments | Length of the study - two years
  The accuracy of the NAP/FE procedure as determined by the discriminant ability of NAP signal in normal or abnormal lung segments, where the reference standard is contemporaneous clinician interpretation of available radiology at the time of study procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Kev Dhaliwal, MRCP PhD, Study Director — University of Edinburgh
Locations (2):
- United Kingdom (2):
  - Ward 118 Intensive Care, Royal Infirmary of Edinburgh, Edinburgh, Edinburgh City
  - Western General Hospital, Edinburgh, Edinburgh City